CLINICAL TRIAL: NCT04988347
Title: The Effect of Spirulina Platensis on Rebound Dyspeptic Symptoms After Discontinuation of Proton Pump Inhibitors: a Phase 2 Clinical Trial
Brief Title: Spirulina Platensis for PPI Withdrawal
Acronym: SpAReDPPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Fernando Fornari, Professor, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 309/2010
Record Dates: First submitted 2021-07-21; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Gastro Esophageal Reflux Disease; Dyspepsia; Rebound Acid Hypersecretion
Keywords: Gastroesophageal reflux disease; Dyspepsia; Proton Pump Inhibitors; Spirulina platensis
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia

STUDY DESIGN:
Intervention Model Description: Forty-five regular users of PPIs entered in a 28-day run-in phase of pantoprazole 40 mg/day, followed by clinical and endoscopic evaluation. In the absence of large hiatal hernia, peptic ulcer, or moderate to severe reflux esophagitis, patients stopped PPIs and were randomly assigned to receive Spirulina (1.6 g/day) or placebo for 2 months, when evaluation was repeated. Primary outcomes were dyspepsia and typical reflux symptoms (either appearance or maintenance of symptoms > 50% from baseline). Intention-to-treat analysis was applied.
Who Masked: Participant, Investigator
Masking Description: Capsules containing Spirulina and placebo were identical
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirulina (Experimental): Active treatment with Spirulina platensis in capsules containing 530 mg, 1 capsule orally each 8 hours, for 60 days
  Interventions: Combination Product: Spirulina platensis
- Placebo (Placebo Comparator): Placebo in capsules, 1 capsule orally each 8 hours, for 60 days
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Combination Product: Spirulina platensis — Active treatment with Spirulina platensis in capsules containing 530 mg, 1 capsule orally each 8 hours, for 60 days
  Arms: Spirulina
Other: Placebo comparator — Placebo in capsules, 1 capsule orally each 8 hours, for 60 days
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Background: Rebound acid hypersecretion after proton pump inhibitors (PPIs) discontinuation may be accompanied by dyspepsia.

Aim: To assess whether Spirulina platensis, by its anti-inflammatory properties, could minimize rebound symptoms after PPIs withdrawal.

DETAILED DESCRIPTION:
Forty-five regular users of PPIs entered in a 28-day run-in phase of pantoprazole 40 mg/day, followed by clinical and endoscopic evaluation. In the absence of large hiatal hernia, peptic ulcer, or moderate to severe reflux esophagitis, patients stopped PPIs and were randomly assigned to receive Spirulina (1.6 g/day) or placebo for 2 months, when evaluation was repeated. Primary outcomes were dyspepsia and typical reflux symptoms (either appearance or maintenance of symptoms > 50% from baseline). Intention-to-treat analysis was applied.

ELIGIBILITY:
Inclusion Criteria:

* Chronic use of any PPIs, either original brand or generic
* Absence of conditions that contraindicate the cessation of PPIs, such as active or recent peptic ulcer, active or recent upper digestive bleeding, regular use of salicylates or non-steroidal anti-inflammatory drugs, moderate to severe reflux esophagitis, and sliding hiatal hernia greater than 3 cm
* Formal agreement to participate

Exclusion Criteria:

* Uncompensated acute and chronic morbidities
* Gastroesophageal surgery
* Cognitive deficit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with dyspeptic symptoms | 60 days
  Relapse of dyspeptic symptoms after PPIs cessation
Number of participants with typical GERD symptoms | 60 days
  Relapse of typical GERD symptoms

SECONDARY OUTCOMES:
Rate of new endoscopic lesions | 60 days
  Endoscopic lesions in the esophagus, stomach and duodenum, after PPIs cessation
Number of participants with microscopic changes in the stomach | 60 days
  number of participants with new or worsened gastric inflammation after PPIs cessation
Number of participants with side effects | 60 days
  Side effects potentially secondary to Spirulina platensis and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fornari, Professor, Principal Investigator — University of Passo Fundo

REFERENCES:
- [Derived] Gronevalt ATM, Bertolin TE, Forcelini CM, Polletto PHM, Pasetti BW, Graeff DB, Rodriguez R, Fornari F. Spirulina Platensis Attenuates Rebound Dyspeptic Symptoms After Proton Pump Inhibitors' Discontinuation: Phase 2 Placebo-controlled Trial. Altern Ther Health Med. 2024 Feb;30(2):18-24. PMID 38401078